CLINICAL TRIAL: NCT03291977
Title: Interest of Fluorescein in Fluorescence-guided Resection of Gliomas: A Randomized Study
Brief Title: Interest of Fluorescein in Fluorescence-guided Resection of Gliomas (FLEGME)
Acronym: FLEGME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC16_9758_FLEGME
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Glioblastoma, Adult
Keywords: surgery - glioblastoma - fluorescein
MeSH Terms: conditions — Glioblastoma | interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorescein sodique FAURE (Experimental): Fluorescein (Fluorescéine sodique FAURE) will be given intravenously during the induction of the anesthesia
  Interventions: Drug: Fluorescéine Sodique Faure
- White-light surgery (Active Comparator): In the control arm, the surgery will be performed under classical conditions (so-called " white-light " surgery).
  Interventions: Procedure: White-light surgery

INTERVENTIONS:
Drug: Fluorescéine Sodique Faure — Fluorescéine Sodique Faure given intravenously during the induction of the anesthesia, at the dose of 3mg/kg, diluted in 50mL of physiological serum, in 10 minutes.
  Arms: Fluorescein sodique FAURE
Procedure: White-light surgery — The surgery will be performed under classical conditions
  Arms: White-light surgery

SUMMARY:
Fluorescence guidance is a safe and efficient tool for glioblastomas resection. The most widely used technique is based on 5-aminolevulinic acid (5ala), which stains glioblastoma cells through a metabolic abnormality and thus helps in defining tumoral edges through a modified microscope. A multicentric, randomized study comparing 5ala guided surgery with conventional procedures showed that this technique doubles the rate of complete removal on post-operative magnetic resonance imaging (MRI), and increases the 6 months progression-free survival. More recently, fluorescein appeared as an interesting alternative fluorophore for glioblastomas, with a highly reduced cost (2.5 euros versus 1000 euros per dose). However its use remains scarcely studied and its clinical benefit unsure. In that context, the investigators propose a randomized trial comparing conventional " white light " surgery with fluorescein-guided resection of glioblastomas, in order to assess the relevance of this technique in glioblastomas removal.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 79
* Karnofsky index > 70 %
* Brain MRI showing a parenchymal lesion with typical features of glioblastoma, < 1week
* Achievable gross total removal, as assessed by the neurosurgical staff
* Written consent

Exclusion Criteria:

* Contraindication to fluorescein
* Contraindication to MRI
* History of brain surgery <6 months
* Guardianship, tutelage or deprivation of liberty
* Pregnancy or breastfeeding
* Participation to other interventional clinical studies

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Gross total removal rates | under 72 hours post-op
  assessed by the absence of residual contrast enhancement on early post-operative MRI

SECONDARY OUTCOMES:
Absolute volumes of tumor remnants | under 72 hours post-op
  assessed in cm3 on early post-operative MRI
Relative volumes of tumor remnants | under 72 hours post-op
  assessed in % on early post-operative MRI
Occurrence of new neurological deficits | under 72 hours post-op
  assessed by the NIHSS
Occurrence of anaphylactic events related to the administration of fluorescein | under 72 hours post-op

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean LE RESTE, Dr, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No